CLINICAL TRIAL: NCT02817542
Title: Trhombus Aspiration in Hyperglycemic ST-elevation myocardiAl InfarcTIon (STEMI) Patients: 1-year Follow-up of the Prospective Randomised TAHITI Study
Brief Title: Trhombus Aspiration in Hyperglycemic ST-elevation myocardiAl InfarcTIon
Acronym: TAHITI
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, Internal medicine full professor, University of Campania Luigi Vanvitelli
Other Study IDs: TAHITI
Record Dates: First submitted 2016-04-28; First posted 2016-06-29 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI TA hyperglycemic subjects: STEMI hyperglycemic patients, percutaneous coronary intervention with TA
  Interventions: Device: percutaneous coronary intervention
- STEMI without TA hyperglycemic subjects: STEMI hyperglycemic patients, percutaneous coronary intervention without TA
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — Percutaneous coronary intervention. Procedures include: Implantation of stents The thrombus aspiration (TA) will be started before crossing the coronary atherosclerosis lesion. A minimum of two syringes (40 mL) of aspirate will be recommended. The guide catheter will be engaged with the coronary ostia when removing the thrombectomy catheter. The guide catheter will be aspirated after thrombectomy to avoid embolisation of air or thrombus. PCI procedure will be done without thrombectomy as per the investigator. Direct stenting will not be mandated in either treatment group. Bailout thrombectomy will be allowed after a failure of the initial PCI alone strategy. The decision about bailout thrombectomy will be made by the interventional cardiologist performing the initial PCI.

SUMMARY:
Background. Patients with ST-Elevation Myocardial Infarction (STEMI) and hyperglycemia on admission have high rates of mortality (1). The management of hyperglycemic patients during STEMI is unclear. We evaluate whether the thrombus aspiration (TA) before primary percutaneous coronary intervention (PCI) may improve STEMI outcomes in hyperglycemic patients (2).

Research Design and Methods. Consecutive 990 hyperglycemic patients with first STEMI undergoing quantitative coronary angiography were studied. Patients were categorized in two groups, either treated by thrombus aspiration v/s patients treated without thrombus aspiration. After discharge from the hospital, all patients will be managed and followed quarterly for 12 months month after event, as outpatients, to perform clinical evaluation, routine analyses and cardiovascular evaluation. The cardiovascular endpoint collected in both cohorts will include cardiac mortality, all-cause mortality and hospitalization for coronary disease and heart failure.

Conclusions. We will attend improved outcomes in hyperglycemic patients treated by the TA before PCI, as compared to hyperglycemic patients treated only by PCI.

DETAILED DESCRIPTION:
The data analyzed in this study will be obtained from hyperglycemic STEMI patients who underwent primary PCI at the Department of Cardiology of the Cardarelli Hospital in Naples Italy between June 1, 2016, and December 1, 2017. This will be a prospective study to compare two therapeutic strategies: PCI plus thrombus aspiration (TA) versus PCI alone in patients with STEMI and hyperglycemia. According to the recent statement by the American Heart Association, hyperglycemia will be defined as an admission plasma glucose level of >140 mg/dl. Inclusion criteria will include: age of 18 years or greater, presentation to the cardiac catheterization laboratory for PCI in the setting of first STEMI, admission plasma glucose level of >140 mg/dl. All STEMI patients will be referred to the cardiac catheterization laboratory within 12 h of presentation. Patients with left ventricular ejection fraction less than 25%, with previous myocardial infarction or previous PCI or/and coronary by-pass grafting, or had received fibrinolytic therapy will be excluded from the study. The following patients will be referred for urgent invasive diagnostics with the intention of performing PCI: symptom duration of 12 hours or less and ST-segment elevation of 0.1 mV or greater in at least 2 contiguous leads (≥0.2 mV in V1-V3) or presumed new-onset left bundle-branch block. The investigation will be conformed with the principles outlined in the Declaration of Helsinki for use of human tissue or subjects. The Institutional Review Board will approve the protocol.

Outcomes The primary outcome of the THAITI study will be all-cause mortality, cardiovascular deaths, recurrent myocardial infarction, cardiogenic shock, and class IV heart failure within 360 days. Other outcomes will include target vessel revascularisation, stent thrombosis, stroke, and transient ischaemic attack within 360 days.

ELIGIBILITY:
Inclusion Criteria:

- age of 18 years or greater, presentation to the cardiac catheterization laboratory for PCI in the setting of first STEMI, admission plasma glucose level ( >140 mg/dl in hyperglycemic Group).

Exclusion Criteria:

- patients with left ventricular ejection fraction less than 25%, with previous myocardial infarction or previous PCI or/and coronary by-pass grafting.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will analyze the consecutive patients presenting with acute myocardial infarction and ST segment elevation (STEMI) admitted to the Department of Cardiology of the Cardarelli Hospital in Naples, Italy. Inclusion criteria will include: age of 18 years or greater, presentation to the cardiac catheterization laboratory for PCI in the setting of first STEMI, admission plasma glucose level ( >140 mg/dl in hyperglycemic Group). All STEMI patients will be referred to the cardiac catheterization laboratory within 12 h of presentation. Patients with left ventricular ejection fraction less than 25%, with previous myocardial infarction or previous PCI or/and coronary by-pass grafting will be excluded.
Sampling Method: Probability Sample
Enrollment: 990 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
cardiovascular death | 12 months
  death caused by loss of heart function such as sudden cardiac arrest or heart attack (myocardial infarction). ECG and cardiac damage markers
recurrent myocardial infarction | 12 months
  Myocardial infarction when there is a blockage in one or more of the arteries to the heart, preventing the heart from receiving enough oxygen-rich blood. If the oxygen in the blood cannot reach the heart muscle, the heart becomes damaged. ECG and cardiac damage markers
heart failure. | 12 months
  Heart failure develops when the heart, via an abnormality of cardiac function (detectable or not), fails to pump blood at a rate commensurate with the requirements of the metabolizing tissues or is able to do so only with an elevated diastolic filling pressure. ECG and echocardiography
acute coronary syndrome | 12 months
  non-ST-elevation acute coronary syndromes (ACSs) and unstable angina. ECG and cardiac damage markers

SECONDARY OUTCOMES:
Target vessel revascularisation | 12 months
  Target lesion revascularization was defined as either repeat percutaneous or surgical revascularization for a lesion anywhere within the stent or the 5-mm borders proximal or distal to the stent. Target lesion revascularization was considered to be ischemia-driven if the target lesion diameter stenosis was ≥50% by quantitative analysis with either electrocardiographic changes at rest or a positive functional study in the distribution of the target lesion, or ≥70% with recurrent symptoms only. Angiography study
stent thrombosis, | 12 months
  Definite or confirmed event with symptoms suggestive of an acute coronary syndrome and angiographic or pathologic confirmation of stent thrombosis.Angiography study
stroke | 12 months
  The sudden death of brain cells due to lack of oxygen, caused by blockage of blood flow or rupture of an artery to the brain. Symptoms: Sudden loss of speech, weakness, or paralysis of one side of the body. CAT scans
transient ischaemic attack | 12 months
  .A transient ischemic attack (TIA) is like a stroke, producing similar symptoms, but usually lasting only a few minutes and causing no permanent damage.CAT scans

CONTACTS AND LOCATIONS:
Overall Officials: Celestino Sardu, MD, PHD, Study Director — University of Campania Luigi Vanvitelli
Locations (1):
- Cardarelli Hospital, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Monthly for 1 year

REFERENCES:
- [Result] Jones DA, Rathod KS, Gallagher S, Jain AK, Kalra SS, Lim P, Crake T, Ozkor M, Rakhit R, Knight CJ, Iqbal MB, Dalby MC, Malik IS, Whitbread M, Mathur A, Redwood S, MacCarthy PA, Weerackody R, Wragg A. Manual Thrombus Aspiration Is Not Associated With Reduced Mortality in Patients Treated With Primary Percutaneous Coronary Intervention: An Observational Study of 10,929 Patients With ST-Segment Elevation Myocardial Infarction From the London Heart Attack Group. JACC Cardiovasc Interv. 2015 Apr 20;8(4):575-84. doi: 10.1016/j.jcin.2014.11.021. PMID 25907084
- [Result] Deedwania P, Kosiborod M, Barrett E, Ceriello A, Isley W, Mazzone T, Raskin P; American Heart Association Diabetes Committee of the Council on Nutrition, Physical Activity, and Metabolism. Hyperglycemia and acute coronary syndrome: a scientific statement from the American Heart Association Diabetes Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2008 Mar 25;117(12):1610-9. doi: 10.1161/CIRCULATIONAHA.107.188629. Epub 2008 Feb 25. PMID 18299505
- [Result] Tilsted HH, Olivecrona GK. To Aspirate or Not to Aspirate: That Is the Question. JACC Cardiovasc Interv. 2015 Apr 20;8(4):585-7. doi: 10.1016/j.jcin.2015.01.014. No abstract available. PMID 25907085
- [Derived] Sardu C, Barbieri M, Balestrieri ML, Siniscalchi M, Paolisso P, Calabro P, Minicucci F, Signoriello G, Portoghese M, Mone P, D'Andrea D, Gragnano F, Bellis A, Mauro C, Paolisso G, Rizzo MR, Marfella R. Thrombus aspiration in hyperglycemic ST-elevation myocardial infarction (STEMI) patients: clinical outcomes at 1-year follow-up. Cardiovasc Diabetol. 2018 Nov 29;17(1):152. doi: 10.1186/s12933-018-0795-8. PMID 30497513